CLINICAL TRIAL: NCT06144970
Title: A Phase I, Double-blind, Randomized, Sham-controlled, Dose-response, Study Evaluating the Safety and Tolerability of TG-C in Subjects with Chronic Discogenic Lumbar Back Pain Due to Degenerative Disc Disease At 6 and 12 Months
Brief Title: Study to Determine the Safety and Tolerability of TG-C in Subjects with Back Pain Due to Degenerative Disc Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kolon TissueGene, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TGC-DDD-101
Record Dates: First submitted 2023-10-31; First posted 2023-11-22 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Degenerative Disc Disease
Keywords: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active Treatment 1 (Active Comparator): Low dose TG-C 1.5 x 10e6 cells
  Interventions: Biological: TG-C Low Dose
- Active Treatment 2 (Active Comparator): Middle dose TG-C 5.0 x 10e6 cells
  Interventions: Biological: TG-C Mid Dose
- Active Treatment 3 (Active Comparator): High dose TG-C 1.5 x 10e7 cells
  Interventions: Biological: TG-C High Dose
- Sham Control (Sham Comparator): single subcutaneous injection of normal saline
  Interventions: Biological: Sham Control

INTERVENTIONS:
Biological: TG-C High Dose — High Dose - 1 mL of the combined TG-C cells
  Arms: Active Treatment 3
Biological: TG-C Mid Dose — Middle Dose - A volume of 2 mL CS10 and 1 mL combined TG-C cells. 1.0 mL volume of the mixed TG-C cells is injected
  Arms: Active Treatment 2
Biological: TG-C Low Dose — Low Dose - A volume of 9 mL CS10 and 1 mL combined TG-C cells. 1.0 mL volume of the mixed TG-C cells is injected
  Arms: Active Treatment 1
Biological: Sham Control — Single subcutaneous injection of normal saline
  Arms: Sham Control

SUMMARY:
The goal of this study is to evaluate the safety and tolerability of TG-C in subjects with chronic discogenic lumbar back pain due to degenerative disc disease. Participants will be administered a single intradiscal injection or subcutaneous injection for sham and followed up with in-clinic visits and telephone calls for 24 months.

DETAILED DESCRIPTION:
A Phase I, Double-blind, Randomized, Sham-controlled, Dose-response, Study Evaluating the Safety and Tolerability of TG-C in Subjects with Chronic Discogenic Lumbar Back Pain due to Degenerative Disc Disease at 6 and 12 Months, male or female subjects with chronic discogenic lumbar back pain due to degenerative disc disease at one level. TG-C is to be administered by a single intradiscal injection to the damaged disc via fluoroscopic guidance. Sham will be a normal saline subcutaneous injection. Subjects will be followed for 24 months with in-clinic visits and telephone calls after study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of >= 22 and <= 70
* Provides written informed consent before undergoing any study specific procedures
* Chronic lower back pain for at least 6 months. Back pain twice as great as leg pain measured using NRS
* VAS between >= 40 and <= 90
* ODI Index >30 and <= 80
* Inadequate response to at least one medication (e.g., NSAID, acetaminophen, muscle relaxant) and some form of formal physical therapy over a period of at least 6 months, within 6-9 months of screening.
* Diagnosis of DDD from L1 to S1, confirmed by patient history and radiographic studies
* Modified Pfirrmann score of 3-7 on MRI
* With or without contained disc herniations of <3 mm protrusion
* If more than 1 degenerative disc is identified. PD must be performed 30 days prior and ensure only one level is the pain generator
* BMI >15 and < 30 kg/m2
* Use birth control

Exclusion Criteria:

* Co-morbid medical condition of the spine or upper extremities
* Grade 2 or higher spondylolisthesis and type III Modic changes around target disc
* Suspicion of full thickness annular tear at disc
* History of endocrine or metabolic disorder
* Rheumatoid or psoriatic arthritis
* Compressive pathology due to stenosis or herniated or sequestered discs
* Symptomatic involvement of more than one lumber disc
* Intact disc bulge/protrusion at >3 mm
* Lumbar intervertebral foraminal stenosis
* Previous surgery at the target disc level
* Epidural or facet joint steroid, platelet rich plasma (PRP) or bone marrow concentrate (BMC) injections, or radio frequency ablation (RFA), within 6 months prior to baseline.
* Pregnant
* Presence of ferromagnetic implants
* Involved in current or pending spinal litigations
* Care is provided under a Worker's Compensation claim
* Physical or mental conditions
* 3 or more of the 5 Waddell signs
* Positive screen for HIV
* Immediate family member of other participating patients
* Participated within 3 months or is concurrently enrolled in non-interventional research
* Transient or has a history of any substance use disorder
* Currently incarcerated
* Investigator site personnel or immediate family or sponsor employee
* On chronic anti-coagulation therapy or have confirmed coagulopathy
* Tested positive on RCR testing at screening

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | 6 and 12 months
  The safety and tolerability of the TG-C injection for the treatment of degenerative disc disease resulting in chronic discogenic lumbar back pain will be evaluated by summarizing adverse events by treatment

SECONDARY OUTCOMES:
Compare pain severity using a Visual Analogue Scale | 6 and 12 months
  Assessment of change from baseline in target back pain using the Visual Analog Scale (VAS). The VAS is a method for the assessment of the intensity of pain. The VAS is a horizontal line, 100 mm in length and anchored by word descriptors at each end (no pain, very severe pain). The patient marks on the line at the point that represents their current state. The VAS score is determined by measuring in millimeters from the left hand end to the point of the mark. The score ranges from "0" or no pain to "100" very severe pain.
Oswestry Disability Index survey | 6 and 12 months
  Survey results compared to patient baseline

OTHER OUTCOMES:
Treatment-emergent adverse events | 18 and 24 months
  The safety and tolerability of the TG-C injection for the treatment of degenerative disc disease resulting in chronic discogenic lumbar back pain will be evaluated by summarizing adverse events by treatment
Compare pain severity using a Visual Analogue Scale | 18 and 24 months
  Assessment of change from baseline in target back pain using the Visual Analog Scale (VAS). The VAS is a method for the assessment of the intensity of pain. The VAS is a horizontal line, 100 mm in length and anchored by word descriptors at each end (no pain, very severe pain). The patient marks on the line at the point that represents their current state. The VAS score is determined by measuring in millimeters from the left hand end to the point of the mark. The score ranges from "0" or no pain to "100" very severe pain.
Oswestry Disability Index survey | 18 and 24 months
  Survey results compared to patient baseline
Numerical Rating Scale | 6, 12, 18, and 24 months
  Compare severity of lower back pain to patient baseline using a Numerical Rating Scale (NRS). Patients rate their pain at baseline and 6 and 12 months after treatment. Patients will use an eleven point numerical scale to record their pain severity with 0 being no pain and 10 being worst possible pain.
Patient Global Impression of Changes | 6, 12, 18, and 24 months
  Patient Global Impression of Changes (PGI-C) is a 7 point scale depicting a patient's rating of overall improvement and their belief about the efficacy of treatment. The score ranges from 1 (very much worse) to 7 (very much improved)
Patient-Reported Outcomes Measurement Information System | 6, 12, 18, and 24 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) is a way to measure patient-reported outcomes (PROs), such as pain, fatigue, physical functioning, emotional distress, and social role participation that have a major impact on quality-of-life. Here patients will answer a survey that consists of 16 questions that measure their physical functions after treatment. Patients will use a 5 point scale to answer the survey questions, with 1 being unable to do and 5 being without any difficulty.
MRI Assessment of Structural Changes of the Spine | 1, 6, 12, and 24 months
  Magnetic Resonance Imaging (MRI) of the lumbar spine will be performed using a 1.5 or 3T MRI machine. The modified Pfirrmann grading system will be used to evaluate MRI signals from the nucleus and inner annular fibers. The modified Pfirrmann grading scale will be used for MRI interpretation. The grading scale uses 8 grades with 1 being uniformly hyperintense and 8 being hyperintense. MRI results will be assessed at 6 and 12 months to observe structural changes to the spine.

CONTACTS AND LOCATIONS:
Overall Officials: Moon Jong Noh, PhD, Study Chair — Kolon TissueGene

IPD SHARING:
Plan to Share IPD: No